CLINICAL TRIAL: NCT01520090
Title: Egyptian Women Knowledge and Use of Different Contraceptive Methods
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, rania mohamed abd el-moez, dr., Ain Shams University
Other Study IDs: 2412012
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2012-01

CONDITIONS: Contraception
Keywords: contraception; family planning; egyptian; knowledge

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Starting from Jan 2012 for an interval of 4 months with minimum number of 1200 egyptian women will be asked to complete a questionairre to evaluate their knowledge of different contraceptive methods

DETAILED DESCRIPTION:
PATIENTS AND METHODS

Sample size, Time of the study:

Starting from Jan 2012 for an interval of 4 months with minimum number of 1200women .

Type of the study:

Analytical crossectional study

Place of the study:

Ain Shams University Hospital, Gynecological outpatient clinic and Amireya primary care medical center (family planning clinic).

Statistical methodology:

SPSS program will be used for data analysis. Appropriate significance tests will be used according to type of data.

After an oral consent is taken from them, Women will be asked to complete a short written questionnaire that includes social data, reproductive information, and some questions about common contraceptive methods.

Testing readability and comprehension of the questionnaire will be done first by collecting 50 questionnaires and analyzing the data.

AIM OF THE WORK The aim of this study is to evaluate knowledge and use of different available contraceptive methods among women attending Ain Shams University maternity hospital in the gynecological outpatient clinic and Amireya primary care medical center (family planning clinic).

ELIGIBILITY:
Inclusion Criteria:

1. Age : 18 -51 years old
2. Using a contraceptive method for at least 6 months continuously.

Exclusion Criteria:

1. Infertile
2. Vaginal bleeding of unknown etiology.
3. Current pregnancy
4. Menopausal

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: egyptian women ,18 -51 years old Using a contraceptive method for at least 6 months continuously.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-03 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
knowledge of the different contraceptive methods | march 2012
  subjects answer the questionairre correctly or at least 70% right answers

SECONDARY OUTCOMES:
correct use of different contraceptive methods | march 2012
  assessing that the subjects use contraceptive methods in correct way based on their knowledge

CONTACTS AND LOCATIONS:
Overall Officials: rania m abdelmoez, M.B., B.CH., Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Maternity Hospital Out-Patient Clinic, Cairo, Egypt